CLINICAL TRIAL: NCT03388658
Title: Safety and Efficacy of Cryoballoon Pulmonary Vein Isolation : a Single Center Registry
Acronym: Gr-CryoFS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.216
Record Dates: First submitted 2017-10-20; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Cryoballoon; Ablation;
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to assess the long-term success rates of pulmonary vein isolation using first and second generation cryoballoons in patients with paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
The success of ablation is determined by the absence of recurrence of atrial fibrillation in the short term beyond 3 months, medium and long term on regular clinical follow-up and ECG holters. The patient cohort followed since 2007 allows a very long-term follow-up of patients who have benefited from atrial fibrillation cryoablation.

Isolation of the pulmonary veins by cryoballoon (IVP) has emerged as an alternative to radiofrequency in the treatment of drug resistant atrial fibrillation (AF). (1) The potential benefits of cryoablation include shorter procedure times, decreased fluoroscopy time, shorter hospital duration, a different rate and type of complications compared to radio frequency offers potential benefits, including Including shorter procedure times, a decrease in the length of hospital stay 1 and a reduction in fluoroscopic time. (2) Effectiveness on a one year follow-up in cryoablation for AF is comparable to that of radiofrequency ablation in a prospective, randomized study with a lower major complication rate (3,4). The number of subjects is limited and most retrospective studies on cryoablation have a limited number of patients or an average follow-up not exceeding one year.

Study of the data and results of the procedures of ablation of AF by cryoablation and long-term follow-up of the patients of the CHU of Grenoble.

Regular monocentric cohort study based on collected data To identify the success rate of cryoablation ablation in paroxysmal and persistent AF

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for ablation of atrial fibrillation at the CHU of Grenoble since the use of this technique (November 2007) until November 2016:
* Paroxysmal atrial fibrillation resistant to antiarrhythmic treatment.
* Persistent atrial fibrillation.
* Patients ≥18 years
* Patients with discernment who signed consent for information on the ablation procedure before surgery.

Exclusion Criteria:

* patient less than 18 years old
* patient who refused to sign informed consent for the procedure of ablation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who have benefited from atrial fibrillation cryoablation in the grenoble University Hospital
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Long term efficacy of cryoballoon ablation for atrial fibrillation (AF) | in a 8-year follow-up period
  Absence of recurrence (recurrence was defined as symptomatic or documented arrhythmia episode of>30 seconds excluding a 3-month blanking period)

SECONDARY OUTCOMES:
Post procedure morbidities | in a 8-year follow-up period
  The secondary outcomes include adverse events related to the procedure: death from any causes, atrial-oesophageal fistula, pericardial tamponade, neurological complication, phrenic nerve palsy, hematoma and vascular complications.
Cryoballoon 1 versus cryoballoon 2 | in a 1200-day follow-up period
  Comparison of acute and long term efficacy in of the first versus second generation cryoballoon
  -The success rate is evaluated at clinical follow-up and Holter, the efficacy of treatment is evaluated by per-ablation data. Total procedure times, catheter time in the left atrium, fluoroscopy time, cryoablation time are collected during the procedure and will be retrospectively analyzed with patient records and ablation records. The comparison will be made on the patient group having been treated with the new techniques and in particular the second generation balloon and those having been treated with the first generation balloon.
Clinical characteristics and predictive factors for success / complications | in a 8-year follow-up period
  The clinical characteristics collected prospectively on the basis since 2007 will be analyzed retrospectively to evaluate one or more factors predicting success or complications of the procedure
Continuation of medical treatment post ablation | in a 1200-day follow-up period
  Continuation of anti-coagulant or anti-arrhythmic treatments beyond 3 months after the procedure will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine VENIER, Dr, Principal Investigator — UniversityHospital Grenoble
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jourda F, Providencia R, Marijon E, Bouzeman A, Hireche H, Khoueiry Z, Cardin C, Combes N, Combes S, Boveda S, Albenque JP. Contact-force guided radiofrequency vs. second-generation balloon cryotherapy for pulmonary vein isolation in patients with paroxysmal atrial fibrillation-a prospective evaluation. Europace. 2015 Feb;17(2):225-31. doi: 10.1093/europace/euu215. Epub 2014 Sep 3. PMID 25186456
- [Background] Cardoso R, Mendirichaga R, Fernandes G, Healy C, Lambrakos LK, Viles-Gonzalez JF, Goldberger JJ, Mitrani RD. Cryoballoon versus Radiofrequency Catheter Ablation in Atrial Fibrillation: A Meta-Analysis. J Cardiovasc Electrophysiol. 2016 Oct;27(10):1151-1159. doi: 10.1111/jce.13047. Epub 2016 Aug 16. PMID 27422848
- [Background] Jiang J, Li J, Zhong G, Jiang J. Efficacy and safety of the second-generation cryoballoons versus radiofrequency ablation for the treatment of paroxysmal atrial fibrillation: a systematic review and meta-analysis. J Interv Card Electrophysiol. 2017 Jan;48(1):69-79. doi: 10.1007/s10840-016-0191-9. Epub 2016 Sep 28. PMID 27683062
- [Background] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Background] Lemes C, Wissner E, Lin T, Mathew S, Deiss S, Rillig A, Heeger C, Wohlmuth P, Reissmann B, Tilz R, Ouyang F, Kuck KH, Metzner A. One-year clinical outcome after pulmonary vein isolation in persistent atrial fibrillation using the second-generation 28 mm cryoballoon: a retrospective analysis. Europace. 2016 Feb;18(2):201-5. doi: 10.1093/europace/euv092. Epub 2015 May 19. PMID 25995389